CLINICAL TRIAL: NCT00630344
Title: A Phase II Trial of RAD001 and Bicalutamide for Androgen Independent Prostate Cancer
Brief Title: RAD001 and Bicalutamide for Androgen Independent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Mary-Ellen Taplin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-316
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer
Keywords: RAD001; bicalutamide; androgen independent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Everolimus; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RAD001 + Bicalutamide (Experimental): RAD001: once daily dose of 10 mg (5 mg tablets)
  Bicalutamide: once daily dose of 50 mg (50 mg tablets)
  1 cycle=28 days
  Both agents are administered continuously until progression of disease or unacceptable toxicity.
  Interventions: Drug: RAD001; Drug: Bicalutamide

INTERVENTIONS:
Drug: RAD001
  Other Names: everolimus
Drug: Bicalutamide
  Other Names: Casodex

SUMMARY:
In the treatment of castration-resistant prostate cancer (CRPC), therapies will long response durations remain elusive as a result of the inherent ability of prostate cancer cells to develop iterative resistance. The goal of this study is to learn if the study drug RAD001 together with Bicalutamide can slow the growth of prostate cancer. The safety of the combination will also be studied.

DETAILED DESCRIPTION:
Bicalutamide, an androgen receptor (AR) antagonist, is frequently used as the first 'secondary hormonal therapy' in combination with another established agent (LHRH: luteinizing hormone-releasing hormone agonist/antagonist) to treat CRPC. A series of studies have shown that RAD001 through inhibition of mammalian target of rapamycin (mTOR) pathway has antitumor and anti-angiogenic activities. The hypothesis is that the combination of an antiandrogen and mTOR inhibitor would have additive and clinically significant effects in CRPC.

STATISTICAL CONSIDERATIONS:

The regimen will be considered promising if the rate of response/favorable outcome is 40% or greater. A rate of 20% (similar to that observed for bicalutamide alone) will not be considered worthy of further study. 38 patients (of whom 36 are assumed to be eligible) will be accrued to the study. If 11 or more patients have a favorable outcome (stable disease > 6 months or response), the combination will be considered worthy of further study. Given this design, there is a 9% probability of declaring the combination effective if the true favorable outcome rate is 20% and a 91% probability of declaring the combination effective if the true favorable outcome rate is 40%.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically documented prostate cancer
* Castration resistant prostate cancer defined as two rising PSAs on castration therapy
* Baseline PSA of 2ns/mL or greater
* Testosterone of 50ng/mL or less
* Patients on LHRH agonist/antagonist must continue therapy at the recommended dosing intervals
* Prior bicalutamide is allowed as long as treatment was for 6 months or longer
* Metastatic disease is not required
* Minimum of four weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy
* ECOG Performance Status equal to or less than 2
* Adequate bone marrow and liver function as outlined by parameters in the protocol

Exclusion Criteria:

* Prior treatment with any investigational drug within the preceding 4 weeks
* Prior treatment with an mTOR inhibitor
* Fasting lipids over the parameters outlined in the protocol
* Chronic treatment with systemic steroids or another immunosuppressive agent
* Patients should not receive immunization with attenuated live vaccines during study period or within one week of study entry
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Other malignancies within the past 3 years except for adequately treated or basal squamous cell carcinomas of the skin
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* Known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001
* Patients with an active, bleeding diathesis or on oral anti-vitamin K medication (except low dose coumarin)
* Men able to conceive and unwilling to practice an effective method of birth control
* Known hypersensitivity to RAD001 or other rapamycins or to its excipients
* History of noncompliance to medical regimens

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Study Chair — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nakabayashi M, Werner L, Courtney KD, Buckle G, Oh WK, Bubley GJ, Hayes JH, Weckstein D, Elfiky A, Sims DM, Kantoff PW, Taplin ME. Phase II trial of RAD001 and bicalutamide for castration-resistant prostate cancer. BJU Int. 2012 Dec;110(11):1729-35. doi: 10.1111/j.1464-410X.2012.11456.x. Epub 2012 Aug 29. PMID 22928480

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RAD001 + Bicalutamide
Started | 36
Completed | 0
Not Completed | 36
Not completed — Adverse Event | 5
Not completed — Progressive Disease | 19
Not completed — Physician Decision | 9
Not completed — Withdrawal by Subject | 1
Not completed — Intercurrent Illness | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Groups:
- RAD-001 in Combination With Bicalutamide: RAD001: once daily dose of 10 mg (5 mg tablets)
  Bicalutamide: once daily dose of 50 mg (50 mg tablets)
  1 cycle=28 days
  Both agents are administered continuously until progression of disease or unacceptable toxicity.
Arm/Group | RAD-001 in Combination With Bicalutamide
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [60 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate is the percentage of patients achieving response taking into consideration measurable disease, bone metastases, and PSA. PSA declines in the absence of both measurable disease and the appearance of new bone lesions or a response in measurable disease without an increase in PSA or the appearance of new bone lesions. Patients with stable disease (SD) lasting at least 6 months will also be considered responders.
  Per RECIST guidelines, for target lesions, complete response (CR) is complete disappearance of all target lesions and partial response (PR) is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. CR or PR confirmation is required within 4 weeks. Per modified PSAWG2 criteria (Scher H, Halabi S, Tannock I et al. JCO 2008) PSA response is defined as PSA decline ≥ 50% from baseline confirmed by a second measurement at least 4 weeks later.
Time Frame: PSA was measured monthly and measurable disease on imaging assessed every 2 cycles in first 8 weeks and every 3 cycles thereafter. In this study cohort, patients were followed on treatment up to approximately 1 year.
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (90% Confidence Interval); unit: percentage of patients
Groups:
- RAD-001 + Bicalutamide: RAD001: once daily dose of 10 mg (5 mg tablets)
  Bicalutamide: once daily dose of 50 mg (50 mg tablets)
  1 cycle=28 days
  Both agents are administered continuously until progression of disease or unacceptable toxicity.
Arm/Group | RAD-001 + Bicalutamide
Number analyzed (Participants) | 36
percentage of patients | 6 [1 to 16]

2. Secondary Outcome: Incidence of Grade 4 Treatment-Related Toxicity
Description: All grade 4 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv3 as reported on case report forms were counted. Incidence is the number of patients experiencing at least one treatment-related grade 4 AE of any type during the time of observation.
Time Frame: Assessed each cycle during therapy and up to 30 days post-therapy completion which is approximately 1 year for patients in this study cohort.
Population: The analysis dataset is comprised of all treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | RAD001 + Bicalutamide
Number analyzed (Participants) | 36
Participants | 0

3. Secondary Outcome: Incidence of Grade 1-3 Treatment-Related Mucositis Toxicity
Description: All grade 1-3 mucositis adverse events (AE) with treatment attribution of possible, probable or definite based on CTCAEv3 as reported on case report forms were counted. Incidence is the number of patients experiencing at least one treatment-related grade 1-3 mucositis AE during the time of observation.
Time Frame: as for outcome 2
Population: The analysis dataset is comprised of all treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | RAD001 + Bicalutamide
Number analyzed (Participants) | 36
Participants | 20

4. Secondary Outcome: Incidence of Grade 1-3 Treatment-Related Rash Toxicity
Description: All grade 1-3 rash adverse events (AE) with treatment attribution of possible, probable or definite based on CTCAEv3 as reported on case report forms were counted. Incidence is the number of patients experiencing at least one treatment-related grade 1-3 rash AE during the time of observation.
Time Frame: as for outcome 2
Population: The analysis dataset is comprised of all treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | RAD001 + Bicalutamide
Number analyzed (Participants) | 36
Participants | 17

5. Secondary Outcome: Incidence of Grade 1-3 Treatment-Related Fatigue Toxicity
Description: All grade 1-3 fatigue adverse events (AE) with treatment attribution of possible, probable or definite based on CTCAEv3 as reported on case report forms were counted. Incidence is the number of patients experiencing at least one treatment-related grade 1-3 fatigue AE during the time of observation.
Time Frame: as for outcome 2
Population: The analysis dataset is comprised of all treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | RAD001 + Bicalutamide
Number analyzed (Participants) | 36
Participants | 16

6. Secondary Outcome: Time to Progression (TTP)
Description: TTP estimated with Kaplan-Meier methods is defined as the time from treatment start to when PSA progression criteria is first met, or the date of measurable or non-measurable disease progression (PD). Absent progression, patients are censored at the date of the last PSA measurement. PSA progression is a ≥25% increase over baseline or nadir PSA, whichever is lowest with a minimum increase of 5 ng/mL. If PSA declines ≥50%, PSA progression is a ≥50% PSA increase above nadir with a minimum increase of 5 ng/mL or back to pretreatment baseline, whichever is lowest. PSA progression requires 2 week confirmation. Per RECIST, PD is at least a 20% increase in sum LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or appearance of new lesions. Non-measurable PD is defined as a worsening bone scan, as indicated by the appearance of two or more new lesions, the appearance of new non-bony metastases or a requirement for radiation therapy.
Time Frame: as for outcome 1
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (Full Range); unit: weeks
Arm/Group | RAD001 + Bicalutamide
Number analyzed (Participants) | 36
weeks | 8.7 [0 to 43.6]

ADVERSE EVENTS:
Time Frame: Assessed each cycle during therapy and up to 30 days post-therapy completion which is approximately 1 year for patients in this study cohort.
Groups:
- RAD-001+ Bicalutamide: RAD001: once daily dose of 10 mg (5 mg tablets)
  Bicalutamide: once daily dose of 50 mg (50 mg tablets)
  1 cycle=28 days
  Both agents are administered continuously until progression of disease or unacceptable toxicity.
Arm/Group | RAD-001+ Bicalutamide
Serious Adverse Events (participants affected / at risk) | 19/36
Other Adverse Events (participants affected / at risk) | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD-001+ Bicalutamide (N=36)
Hemoglobin (Blood and lymphatic system disorders) | 2
Double vision (Eye disorders) | 1
Muco/stomatitis by exam- oral cavity (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Pain-other (General disorders) | 1
Infection neut-anal/perianl (Infections and infestations) | 1
Leukocytes (Investigations) | 1
Alkaline phosphatase (Investigations) | 1
CPK (Investigations) | 1
Creatinine (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Bone-pain (Musculoskeletal and connective tissue disorders) | 1
Neuropathy CN XII tongue (Nervous system disorders) | 1
Speech impairment (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Glomerular filtration rate (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD-001+ Bicalutamide (N=36)
Hemoglobin (Blood and lymphatic system disorders) | 2
Neutrophils (Investigations) | 1
Hematologic-other (Blood and lymphatic system disorders) | 1
Hypotension (Vascular disorders) | 1
Cardiac-other (Cardiac disorders) | 1
Fatigue (General disorders) | 14
Fever w/o neutropenia (General disorders) | 3
Insomnia (Psychiatric disorders) | 3
Rigors/chills (General disorders) | 1
Weight loss (Investigations) | 4
Constitutional- other (General disorders) | 3
Bruising (Injury, poisoning and procedural complications) | 1
Burn (Injury, poisoning and procedural complications) | 1
Chelitis (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 10
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 6
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Skin-other (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 7
Constipation (Gastrointestinal disorders) | 5
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 9
Dry mouth (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Muco/stomatitis by exam- oral cavity (Gastrointestinal disorders) | 10
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 7
Taste disturbance (Nervous system disorders) | 6
Vomiting (Gastrointestinal disorders) | 3
GI-other (Gastrointestinal disorders) | 2
Bladder- hemorrhage (Renal and urinary disorders) | 1
Urinary hemorrhage NOS (Renal and urinary disorders) | 2
Nose- hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Hemorrhage-other (Vascular disorders) | 1
Infection Gr0-2 neut- anal/perianl (Infections and infestations) | 1
Infection Gr0-2 neut- lung (Infections and infestations) | 1
Edema limb (General disorders) | 3
Lymphatics-other (Blood and lymphatic system disorders) | 1
ALT- SGPT (Investigations) | 3
AST- SGOT (Investigations) | 3
Hypercholesterolemia (Investigations) | 3
CPK (Investigations) | 6
Creatinine (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Extremity upper (function) (Musculoskeletal and connective tissue disorders) | 1
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 3
Nonneuropathic facial muscle weak (Nervous system disorders) | 1
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Extrapyramidal movement (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 2
Neuropathy CN VI lateral deviation eye (Nervous system disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 1
Psychosis (Psychiatric disorders) | 1
Tremor (Nervous system disorders) | 1
Dry eye syndrome (Eye disorders) | 1
Double vision (Eye disorders) | 1
Vision-blurred (Eye disorders) | 2
Abdomen- pain (Gastrointestinal disorders) | 1
Back- pain (Musculoskeletal and connective tissue disorders) | 7
Bone- pain (Musculoskeletal and connective tissue disorders) | 2
Buttock- pain (Musculoskeletal and connective tissue disorders) | 1
Chest/thoracic pain NOS (General disorders) | 1
Dental/teeth/peridontal- pain (Gastrointestinal disorders) | 1
Extremity-limb- pain (Musculoskeletal and connective tissue disorders) | 2
Head/headache (Nervous system disorders) | 4
Joint- pain (Musculoskeletal and connective tissue disorders) | 4
Muscle- pain (Musculoskeletal and connective tissue disorders) | 1
Neck- pain (Musculoskeletal and connective tissue disorders) | 2
Oral cavity- pain (Gastrointestinal disorders) | 2
Pain NOS (General disorders) | 2
Pelvic- pain (Reproductive system and breast disorders) | 1
Penis- pain (Reproductive system and breast disorders) | 1
Throat/pharynx/larynx- pain (Respiratory, thoracic and mediastinal disorders) | 3
Pain-other (General disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 2
Cystitis (Renal and urinary disorders) | 1
Obstruction-bladder (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 4
Gynecomastia (Reproductive system and breast disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No